CLINICAL TRIAL: NCT02290951
Title: An Open-Label, Multi-Center Phase 1 Study to Investigate the Safety and Tolerability of REGN1979, an Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody, in Patients With CD20+ B-Cell Malignancies Previously Treated With CD20-Directed Antibody Therapy (ELM-1)
Brief Title: Study to Investigate the Safety and Tolerability of Odronextamab in Patients With CD20+ B-Cell Malignancies
Acronym: ELM-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-HM-1333; 2015-004491-30 (EudraCT Number); 2024-514938-20-00 (EU CTIS Number)
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-08

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Diffuse large B-cell lymphoma (DLBCL); Follicular lymphoma (FL); Aggressive lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): DLBCL post CAR-T
  Interventions: Drug: Odronextamab multiple dose levels
- 1N Part B (Experimental): FL
  Interventions: Drug: Odronextamab multiple dose levels
- 2N Part B (Experimental): DLBCL
  Interventions: Drug: Odronextamab multiple dose levels

INTERVENTIONS:
Drug: Odronextamab multiple dose levels — Administered by intravenous (IV) infusion
  Other Names: REGN1979
  Arms: Part A
Drug: Odronextamab multiple dose levels — Administered by subcutaneous (SC) injection
  Other Names: REGN1979
  Arms: 1N Part B; 2N Part B

SUMMARY:
This study has two parts with distinct study objectives and study design. In part A, odronextamab is studied as an intravenous (IV) administration with a dose escalation and a dose expansion phase for B-NHL and CLL. The dose escalation phase for B-NHL and the CLL study are closed at the time of protocol amendment 17. In part B, odronextamab is studied as a subcutaneous (SC) administration with a dose finding and a dose expansion phase for B-NHL.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have documented CD20+ B-cell malignancy, with active disease not responsive to prior therapy, for whom no standard of care options exists, and for whom treatment with an anti-CD20 antibody may be appropriate:

   * Part A (IV administration) B-NHL confirmed by National Cancer Institute (NCI) working group criteria
   * Part B (SC administration): Confirmed diagnosis of B-NHL requiring therapy as defined by WHO classification 2017
2. Patients with B-NHL must have had prior treatment with an anti-CD20 antibody therapy. Patients with CLL (Part A only) are not required to have received prior treatment with an anti-CD20 antibody therapy as defined in the protocol.

   * For the inclusion in the disease-specific expansion cohort enrolling DLBCL patients after failure of CAR-T therapy, the patient must have recovered from the toxicities of the lymphodepletion therapy and CAR-T infusion.
   * For inclusion in Part B, patients must have FL grade 1-3a or DLBCL (with or without prior CAR-T) per the criteria above, and:
   * Patients with FL grade 1-3a and DLBCL must have received at least 2 prior lines of systemic therapy, including an anti-CD20 antibody and an alkylating agent
3. All patients must have at least one bi-dimensionally measurable lesion ≥1.5 cm) documented by CT or MRI scan, if CT scan is not feasible.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
5. Life expectancy of at least 6 months
6. Adequate bone marrow function as described in the protocol
7. Adequate organ function as described in the protocol
8. Willingness to undergo mandatory tumor biopsy pretreatment, if in the opinion of the investigator, the patient has an accessible lesion that can be biopsied without significant risk to the patient.
9. Willing and able to comply with clinic visits and study-related procedures
10. Provide signed informed consent or legally acceptable representative

Key Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known or suspected CNS involvement by non-primary CNS NHL
2. History of or current relevant CNS pathology such as

   * Epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis, or
   * Evidence for presence of inflammatory lesions and/or vasculitis on cerebral MRI
3. Standard anti-lymphoma chemotherapy (non-biologic) or radiotherapy within 28 days prior to first administration of study drug
4. Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV) infection [(as noted by detectable levels on a blood polymerase chain reaction (PCR) assay)].

   1. Patients with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus deoxyribonucleic acid (DNA) that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted upon consultation with the physician managing the infection.
   2. Patients who show detectable levels of CMV at screening will need to be treated with appropriate antiviral therapy and demonstrate at least 2 undetectable levels of CMV by PCR assay (at least 7 days apart) before being re-considered for eligibility.
5. Patients who have received a live vaccination within 28 days of first dose of study treatment

Note: Other protocol Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Safety/overall frequency of adverse events (AEs) | Up to 24 months
  Part A and B
Safety/dose limiting toxicities (DLTs) | Up to 28 days
  Part A and B
Antitumor activity as measured by the objective response rate (ORR) | Through study completion, an average of 24 months
  Expansion Cohorts:
  • Diffuse large B-cell lymphoma (DLBCL) after failure of CAR-T therapy
  Part A

SECONDARY OUTCOMES:
Pharmacokinetics (Concentration of odronextamab) | Up to 10 months
  Peak plasma concentration (Cmax) of odronextamab
  Part A and B
Incidence of anti-drug antibodies (ADA) to odronextamab | Over time; up to approximately 15 months
  Part A and B
Titer of ADA to odronextamab | Over time; up to approximately 15 months
  Part A and B
Incidence of neutralizing antibodies (NAb) to odronextamab over time | Over time; Up to approximately 15 months
  Part A and B
Objective response rate (ORR) | Through study completion, an average of 24 months
  For dose escalation portion and expansion cohorts:
  * Aggressive lymphoma expansion cohort 2
  * FL grade 1-3a expansion cohorts 1 and 2 (Part A)
  For dose escalation and dose expansion cohorts:
  * FL grade 1-3a
  * DLBCL
  * DLBCL post CAR T failure (Part B)
Progression-free survival | Up to 48 months
  Part A and B
Overall Survival | Until death or lost to follow-up/ withdrawal, approximately up to 48 months
  Part A and B
Duration of response (DOR) | Until progression, approximately up to 48 months
  Part A and B
Minimal residual disease (MRD) for patients with CLL | Up to 24 months
  Part A
Duration of Complete Response (DOCR) | Until progression, approximately up to 48 months
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (22):
- United States (10):
  - University of California, Irvine, Orange, California
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute (Massachusetts General Hospital and Beth Israel), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
- France (3):
  - Centre Henri Becquerel, Rouen, Haute-Normandie
  - CHU Hôpital Lyon Sud, Lyon
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Universitatsklinikum Wurzburg, Würzburg, Bavaria, Germany
- Israel (6):
  - Meir Medical Center, Kfar Saba, Central District
  - The Chaim Sheba Medical Center, Tel-Hashomer, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Assuta Ashdod University Hospital, Ashdod, Southern District
  - Rambam Health Care Campus - Hematology and Bone Marrow Transplantation Institute, Haifa
  - Lady Davis Carmel Medical Center, Haifa
- United Kingdom (2):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Topp MS, Matasar M, Allan JN, Ansell SM, Barnes JA, Arnason JE, Michot JM, Goldschmidt N, O'Brien SM, Abadi U, Avivi I, Cheng Y, Flink DM, Zhu M, Brouwer-Visser J, Chaudhry A, Mohamed H, Ambati S, Crombie JL. Odronextamab monotherapy in R/R DLBCL after progression with CAR T-cell therapy: primary analysis of the ELM-1 study. Blood. 2025 Apr 3;145(14):1498-1509. doi: 10.1182/blood.2024027044. PMID 39786390
- [Derived] Bannerji R, Arnason JE, Advani RH, Brown JR, Allan JN, Ansell SM, Barnes JA, O'Brien SM, Chavez JC, Duell J, Rosenwald A, Crombie JL, Ufkin M, Li J, Zhu M, Ambati SR, Chaudhry A, Lowy I, Topp MS. Odronextamab, a human CD20xCD3 bispecific antibody in patients with CD20-positive B-cell malignancies (ELM-1): results from the relapsed or refractory non-Hodgkin lymphoma cohort in a single-arm, multicentre, phase 1 trial. Lancet Haematol. 2022 May;9(5):e327-e339. doi: 10.1016/S2352-3026(22)00072-2. Epub 2022 Apr 1. PMID 35366963
- [Derived] Zhu M, Olson K, Kirshner JR, Khaksar Toroghi M, Yan H, Haber L, Meagher C, Flink DM, Ambati SR, Davis JD, DiCioccio AT, Smith EJ, Retter MW. Translational findings for odronextamab: From preclinical research to a first-in-human study in patients with CD20+ B-cell malignancies. Clin Transl Sci. 2022 Apr;15(4):954-966. doi: 10.1111/cts.13212. Epub 2022 Jan 7. PMID 34997701